CLINICAL TRIAL: NCT05058846
Title: Pilot Study of Pancreatic Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 209514; NCI-2021-07922 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Endoscopic Ultrasound-Guided Fine Needle Aspiration; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, tissue, and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I: No strong family history of pancreatic cancer: Participants in Group 1 consist of BRCA, ATM and PALB2 mutation carriers without a strong family history of pancreatic cancer and can choose to undergo annual magnetic resonance imaging (MRI)/Magnetic resonance cholangiopancreatography (MRCP) and EUS screening, or they may opt out of annual MRI screening. Participants also have the opportunity to co-enroll in the University of California, San Francisco (UCSF) BRCA Center Biorepository for biospecimen/biomarker collection and will complete surveys, including the optional eGene questionnaire, which involves co-enrollment in the eGene Study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Cholangiopancreatography; Procedure: Magnetic Resonance Imaging; Procedure: Endoscopic ultrasound; Other: Questionnaires
- Group II: Strong family history of pancreatic cancer: Participants in Group 2 consist of BRCA, ATM and PALB2 mutation carriers with a strong family history of pancreatic cancer. Participants may undergo annual MRI/MRCP screening and may also elect to get an endoscopic ultrasound (EUS) every other year. Participants also have the opportunity to co-enroll in the UCSF BRCA Center Biorepository for biospecimen/biomarker collection and will complete surveys, including the optional eGene questionnaire, which involves co-enrollment in the eGene Study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Cholangiopancreatography; Procedure: Magnetic Resonance Imaging; Procedure: Endoscopic ultrasound; Other: Questionnaires

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood, tissue, and saliva collection
  Other Names: Biological Sample Collection
Procedure: Magnetic Resonance Cholangiopancreatography — Undergo MRCP
  Other Names: MRCP
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Endoscopic ultrasound — Undergo endoscopic ultrasound
  Other Names: EUS
Other: Questionnaires — Complete the following questionnaires: Pancreatic Cancer Knowledge Survey, Pancreatic Cancer Worry Scale, Disease Specific Perceived Risk Survey, eGene Questionnaire
  Other Names: Surveys

SUMMARY:
This study investigates how often abnormal findings from routine magnetic resonance imaging occur in people with genetic mutations in BReast CAncer gene. (BRCA), ataxia telangiectasia mutated gene (ATM), or PALB2 screened for pancreatic cancer. This study may lead to a greater understanding of cancer and potentially, improvements in cancer screening and treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the event rate of abnormal magnetic resonance imaging (MRI) and Endoscopic ultrasound (EUS) findings in screened study participants.

SECONDARY OBJECTIVES:

I. To determine the rates of high-grade pancreatic neoplasia precursors (intraductal papillary mucinous neoplasm (IPMN)-high-grade dysplasia (HGD)) and pancreatic intraepithelial neoplasia-3 [PanIN-3]) and pancreatic ductal adenocarcinoma (PDAC) among all study participants.

II. To understand rates of procedures (biopsies and surgeries) among all study participants.

EXPLORATORY OBJECTIVES:

I. To create a biorepository of all participants through the collection of saliva, blood, and tissue, combined with imaging findings and robust clinical annotation of patient health behaviors in all study participants.

II. To explore knowledge, attitudes, and anxiety related to pancreatic cancer screening at annual intervals in all study participants.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: GROUP I: Participants may opt to undergo MRI/magnetic resonance cholangiopancreatography (MRCP) or alternating MRI/MRCP and EUS annually for 10 years or complete questionnaires over 10 minutes and undergo blood, saliva and tissue sample collection.

GROUP II: Participants may undergo MRI/MRCP or alternating MRI/MRCP and EUS annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

Ability to provide consent and willing, and able to comply with study procedures Ability to read and speak English

GROUP I:

* Documentation of pathogenic or likely pathogenic germline BRCA 1 and 2, ATM or PALB2 germline genetic mutation
* No strong family history of pancreatic cancer (defined as having >= 1 first-degree or second-degree relative with a history of pancreatic cancer)
* Age >= 50 years old at time of consent.

GROUP II:

* Documentation of pathogenic or likely pathogenic germline BRCA 1 and 2, ATM, or PALB2 germline genetic mutation
* Has strong family history of pancreatic cancer (defined as having >= 1 first-degree or second-degree relative with a history of pancreatic cancer)
* Age >= 18 years old at time of consent (screening generally begins 10 years prior to the earliest pancreatic cancer in the family)

Exclusion Criteria:

* Prior or active pancreatic cancer.
* Pregnant women are excluded from this study because effects of an MRI on developing fetus is unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with germline BRCA, ATM or PALB2 mutation with or without a strong family history of pancreatic cancer. Eligible participants will be identified through UCSF's Hereditary Cancer Clinic or referred through UCSF's gastroenterology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2032-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with of abnormal magnetic resonance imaging (MRI) findings | Up to 10 years
  Proportion of participants with an abnormal MRI finding will be reported as an event. An estimated event rate of 19% in participants with a strong family history (FH) of pancreatic cancer and 10% in those participants without a strong FH of pancreatic cancer and 95% binomial confidence intervals (CIs) will also be reported.

SECONDARY OUTCOMES:
Overall Cancer Detection Rate | Up to 10 years
  Will estimate and infer 95% binomial confidence intervals (CI) and the overall cancer detection rate for all participants on study.
Rates of high-grade neoplastic precursors | Up to 10 years
  Will estimate and infer 95% binomial CI and the overall rate of high-grade pancreatic neoplasia precursors (IPMN-HGD and PanIN-3) for all participants on study.
Rates of pancreatic ductal adenocarcinoma (PDAC) | Up to 10 years
  Will estimate and infer 95% binomial CI and the overall rate of PDAC for all participants on study.
Proportion of participants who have additional medical procedures | Up to 10 years
  The proportion of participants who have obtained a biopsy or underwent a surgical procedure related to a possible diagnosis of cancer will be reported.

OTHER OUTCOMES:
Scores on the Pancreatic Cancer Knowledge Survey | Baseline, approximately 1 day
  The Pancreatic Cancer Knowledge Survey is a 3-item, multiple choice questionnaire designed to gauge participant knowledge on the risk for pancreatic cancer in patients with inherited cancer risk mutations, specifically pancreatic ductal adenocarcinoma (PDAC) and given to participants at time of enrollment. Scores range from 0 to 3, with a higher score indicating a greater knowledge of general pancreatic cancer information.
Change in scores on the Pancreatic Cancer Worry Scale | Up to 10 years
  The Pancreatic Cancer Worry Scale is a 4-item, multiple choice questionnaire which assesses the participants level of worry about developing or existing pancreatic cancers. Scores for each item range from 1='rarely or never'/'not at all' to 4="All of the time / very concerned" for a total score range of 4-16. Higher scores indicate a greater level of worry.
Change in scores on the Disease Specified Perceived Risk Survey | Up to 10 years
  The Disease Specified Perceived Risk Survey is a 4-item survey which addresses participant's perceived risk of developing cancer. Scores for each item range from 0 to 100, for a total score range of 0-400. Higher scores indicating a greater level of perceived risk.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela N Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No